CLINICAL TRIAL: NCT04571801
Title: Optimization of Sepsis Therapy Based on Patient-specific Digital Precision Diagnostics
Acronym: DigiSep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Noscendo GmbH, Germany (Unknown); Health Economics and Health Care Management, Bielefeld University (Unknown); Institute of Medical Biometry and Informatics, University of Heidelberg (Unknown); Coordination Centre for Clinical Trials (KKS), University of Heidelberg (Unknown); Department of Infectious Diseases, University Hospital Essen (Unknown); Center for Infectious Diseases and Infection Control, Jena University Hospital (Unknown); Department of Anesthesiology, Heidelberg University Hospital (Unknown); AOK Rheinland/Hamburg (Industry); Barmer Health Insurance, Germany (Unknown); Techniker Health Insurance, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DigiSep 01
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Bacteremia; Blood culture; Next generation sequencing; Digital precision diagnostics; Desirability of outcome ranking / response adjusted for duration of antibiotic risk (DOOR/RADAR) score
MeSH Terms: conditions — Sepsis; Shock, Septic; Bacteremia

STUDY DESIGN:
Intervention Model Description: Arm 1: Standard diagnostics (Microbial diagnostics by means of standard culture methods + optional consultation of experts in the field of infectious diseases) within the first 72 h after diagnosis
  Arm 2: Standard diagnostics + NGS (Microbial diagnostics using standard culture methods + Next Generation Sequencing + optional consultation of experts in the field of infectious diseases) within the first 72 h after diagnosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Active Comparator): Standard diagnostics
  Interventions: Diagnostic Test: Standard diagnostics
- 2 (Experimental): Standard diagnostics + NGS
  Interventions: Diagnostic Test: Next Generation Sequencing (NGS)

INTERVENTIONS:
Diagnostic Test: Standard diagnostics — Standard diagnostics (Microbial diagnostics by means of standard culture methods + optional consultation of experts in the field of infectious diseases) within the first 72 h after diagnosis of sepsis / septic shock
  Arms: 1
Diagnostic Test: Next Generation Sequencing (NGS) — Standard diagnostics + NGS (Microbial diagnostics using standard culture methods + Next Generation Sequencing + optional consultation of experts in the field of infectious diseases) within the first 72 h after diagnosis of sepsis / septic shock
  Arms: 2

SUMMARY:
Sepsis is triggered by an infection and represents one of the greatest challenges of modern intensive care medicine. With regard to a targeted antimicrobial treatment strategy, the earliest possible pathogen detection is of crucial importance. Until now, culture-based detection methods represent the diagnostic gold standard, although they are characterized by numerous limitations. Culture-independent molecular diagnostic procedures may represent a promising alternative. In particular, the concept of plasmatic detection of circulating, free DNA employing next-generation sequencing (NGS) has shown to be suitable for the detection of disease-causing pathogens in patients with bloodstream infections.

The DigiSep-Trial is a randomized, controlled, interventional, multicenter trial to characterize the effect of the combination of NGS-based digital precision diagnostics, standard-of-care microbiological analyses and optional expert exchanges compared to solely standard-of-care microbiological analyses in the clinical picture of sepsis / septic shock. The study examines in 410 patients (n = 205 per arm) with sepsis / septic shock whether the so-called DOOR-RADAR (Desirability of Outcome Ranking / Response Adjusted for Duration of Antibiotic Risk) score (representing a combined endpoint including the criteria (1) inpatient admission time, (2) consumption of antibiotics, (3) mortality and (4) acute renal failure (ARF)) can be significantly improved, by application of an additional NGS-based diagnostic concept. We also aim to investigate whether the new diagnostic procedure is cost-effective. It is postulated that the inpatient admission time, mortality rate, incidence of ARF, the duration of antimicrobial therapy as well as the costs of complications and outpatient aftercare can be reduced. Moreover, a significant improvement in the quality of life (QoL) of the affected patients can be expected.

Extensive preparatory work suggests that NGS-based diagnostics have higher specificity and sensitivity compared to standard-of-care microbiological analyses for detecting bloodstream infections. This preliminary work for the DigiSep-Trial with the help of an interventional study design provides the optimal basis to establish this new concept as part of the national standard based on the best possible evidence.

DETAILED DESCRIPTION:
Sepsis is a disease which is triggered by an infection and represents one of the greatest challenges of modern intensive care medicine. With regard to targeted anti-microbial therapy, the earliest possible pathogen detection is of crucial importance. Until now, culture-based detection methods represent the gold standard for diagnosis, although numerous limitations characterize these. In this context, culture-independent molecular biological processes are an alternative. In particular, the concept of serum detection of circulating, free DNA employing next-generation sequencing (NGS) seems to represent a promising diagnostic procedure in patients with bloodstream infections. The applicant's extensive preparatory work suggests that NGS-based diagnostics using the SIQ score have higher specificity and sensitivity compared to traditional culture-based methods for detecting bloodstream infections. This preliminary work for the DigiSep trial with the help of interventional study design provides the optimal basis to establish this new concept as part of the national standard based on the best possible evidence. The DigiSep trial is intended to characterize the effect of the combination of digital precision diagnostics, expert exchange and culture-based standard diagnostics compared to a purely culture-based conventional diagnosis in the clinical picture of sepsis / septic shock. The study examines in 410 patients (n = 205 per arm) with sepsis / septic shock whether the so-called DOOR-RADAR score (Desirability of Outcome Ranking / Response Adjusted for Duration of Antibiotic Risk Score) can be significantly improved, by application of the NGS. We also aim to also study whether the new procedure is cost-effective. It is postulated that the inpatient admission time, mortality rate, incidence of acute renal failure (ARF), the duration of anti-microbial therapy as well as the costs of complications and outpatient aftercare can be reduced. Also, a significant improvement in the quality of life of the affected patients can be expected.

As part of the study, the essential data is collected once at the time of sepsis (= onset). The culture-based diagnostics include the guideline-oriented collection of 2 blood culture sets (2 x aerobic / 2 x anaerobic) to the onset and three days later. At the same time, serum samples are obtained for NGS-based pathogen diagnostics. Additional sampling for NGS-based diagnostics can be made up to day 14 after onset or whenever the attending physician establishes a clinical indication for the collection of further blood cultures. The aforementioned cultures vs NGS-based pathogen diagnostics are also accompanied by extended immunological monitoring from blood plasma samples as well as an NGS-based transcriptome analysis. The associated sampling takes place at the time of onset, 3, 7 and 14 days after the beginning of sepsis. Routine microbiological findings from other biological samples (e.g. surgical swabs, drainage secretions, tracheal secretions, tissue samples) are included in the evaluation if these were collected three days before or after the extraction of serum samples for NGS-based diagnostics. The clinical data collection is also carried out at the time of sepsis (= onset), 3, 7 and 14 days later, analogous to the above-mentioned sample collection. The final outcome evaluation takes place 28 days (= 28 d) after the onset of sepsis. The study-related burden on the individual study patient includes a total of 17 ml of whole blood for NGS-based diagnostics, the four samples of 7.5 ml of whole blood for immunological monitoring and the four samples of 2.7 ml of whole blood for transcriptome analysis. The minimum total volume, therefore, amounts to the collection of approximately 75 ml of whole blood within the first 14 days after the onset of sepsis. The sampling takes place with the collection of the blood cultures or within the framework of the daily routine blood samples so that no further venous punctures are required here. Infection parameters such as procalcitonin (PCT) are carried out within the framework of daily regular blood collection and therefore, do not require any additional vascular punctures. The same principle applies to the collection of blood cultures which are routinely obtained as part of standard diagnostics in patients with suspected or proven sepsis. The required blood samples of two 40 ml of whole blood (each two sets of 2 x aerobic / 2 x anaerobic = 4 x 10 ml = 40 ml) therefore do not represent any additional burden due to the study. A further additional burden for the patient concerning invasive procedures or examinations is not expected in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who develop sepsis or septic shock within < 24 h in accordance with the new sepsis definition (Sepsis-3) in the above-mentioned participating centers and consent to participation in the study will be included.

General inclusion criteria:

* Written consent by the study participant or a legally appointed representative
* Age >18 years

Sepsis:

* Life-threatening organ dysfunction due to a dysregulated immune response on the basis of a suspected or proven infection
* Detection of organ dysfunction indicated by SOFA score of ≥ 2 points Alternative:

Change of the quick (q) SOFA score of 2 points as an indication of a sepsis

Or septic shock:

* Persistent hypotension despite adequate volume substitution, which necessitates the use of vasopressors, to maintain an arterial medium pressure of > 65 mmHg
* Serum lactate > 2 mmol/l (18 mg/dl)

Exclusion Criteria:

* Age < 18 years
* Refusal to participate in the study
* Probable discharge of the patient from the intensive care unit within the first 72 h of initial study inclusion
* Palliative therapy approach
* Death of the patient is already foreseeable or inevitable at trial inclusion
* Patients who have already been included in the study but require re-admission to the intensive care unit cannot be included a second

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking / Response Adjusted for Duration of Antibiotic Risk-Score | 28 days
  DOOR/RADAR-score [points], (min. 1, max. 5), a lower score indicates a better outcome

SECONDARY OUTCOMES:
Disease severity | at 90 and 180 days
  Long term mortality [%]
Disease severity | at 28, 90, and 180 days
  Hospital length of stay [days]
Degree of organ dysfunction/-failure | at 28, 90, and 180 days
  Duration of mechanical ventilation [days]
Degree of organ dysfunction/-failure | during 28 days
  Length of time until shock resolution [hours]
Degree of organ dysfunction/-failure | at 28, 90, and 180 days
  Ongoing need for renal replacement therapy [%]
Microbiological outcome | at 28, 90, and 180 days
  Cumulative need for anti-infective drugs [days]
Microbiological outcome | during 28 days
  Beginning of a targeted anti-infective treatment regimen [days]
Health economic outcome | at 28, 90, and 180 days
  Utilization of healthcare ressources (outpatient and inpatient) [Euro]
Health economic outcome | at 28, 90, and 180 days
  Policyholder costs (outpatient and inpatient) [Euro]
Economic outcome | at 28, 90, and 180 days
  Disease-related absence from work [days]
Quality-of-life (QoL) based on VR-36 questionnaire | 90 and 180 days
  VR-36 questionnaire [points] including 2 summary components, 8 scales, 36 items, a higher score indicates a higher Quality-of-Life (QoL)
Quality-of-life (QoL) based on EQ-5D-5L questionnaire | at 0, 90 and 180 days
  EQ-5D-5L questionnaire [points] including 10 items, a higher score indicates a higher Quality-of-Life (QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Brenner, MD, Principal Investigator — Department of Anesthesiology, University Hospital Essen
Locations (22):
- Germany (22):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Heidenheim Hospital, Heidenheim, Baden-Wurttemberg
  - Konstanz Hospital, Konstanz, Baden-Wurttemberg
  - University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - University Hospital TU München, München, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - University Hospital Würzburg, Würzburg, Bavaria
  - Klinik Evangelisches Krankenhaus Luckau gGmbH, Luckau, Brandenburg
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Helios Dr. Horst Schmidt Hospital, Wiesbaden, Hesse
  - University Hospital Göttingen, Göttingen, Lower Saxony
  - University Hospital Hannover (MHH), Hanover, Lower Saxony
  - University Hospital Rostock, Rostock, Mecklenburg-Vorpommern
  - University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Klinik Evangelisches Krankenhaus Bethel gGmbH Bielefeld, Bielefeld, North Rhine-Westphalia
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Köln, Cologne, North Rhine-Westphalia
  - University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - University Hospital Leipzig, Leipzig, Saxony
  - University Hospital Charité, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Researchers with access to data are limited to the project partners involved. Researchers will receive pseudonymized data sets for data evaluations. A prerequisite for the transfer of the data to the project partners is the written consent of the patients.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Brenner T, Skarabis A, Stevens P, Axnick J, Haug P, Grumaz S, Bruckner T, Luntz S, Witzke O, Pletz MW, Ruprecht TM, Marschall U, Altin S, Greiner W, Berger MM; TIFOnet Critical Care Trials Group. Optimization of sepsis therapy based on patient-specific digital precision diagnostics using next generation sequencing (DigiSep-Trial)-study protocol for a randomized, controlled, interventional, open-label, multicenter trial. Trials. 2021 Oct 18;22(1):714. doi: 10.1186/s13063-021-05667-x. PMID 34663439